CLINICAL TRIAL: NCT05280821
Title: Comparing Oral Iron Supplementation Using Alternate-day Dosing to the Standard of Care Consecutive-day Dosing in Iron-depleted Women With or Without Mild Anemia: a Randomized Controlled Trial in the Philippines
Brief Title: Alternate Day vs. Daily Iron Supplementation in Iron Depleted Women in the Philippines
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: St. Luke's Medical Center (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAPS_PH
Record Dates: First submitted 2022-02-23; First posted 2022-03-15 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and investigators are blinded, double blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consecutive Day Dosing (Active Comparator): This arm will daily receive iron capsules for 3 months, followed by daily placebo capsules for 3 months.
  Interventions: Dietary Supplement: daily ferrous sulfate
- Alternate Day Dosing (Experimental): This arm will receive iron capsules alternating with placebo capsules for 6 months.
  Interventions: Dietary Supplement: alternate day ferrous sulfate

INTERVENTIONS:
Dietary Supplement: daily ferrous sulfate — Daily intake of 100 mg ferrous sulfate capsules for 3 months
  Arms: Consecutive Day Dosing
Dietary Supplement: alternate day ferrous sulfate — Alternate day intake of 100 mg ferrous sulfate capsules for 6 months
  Arms: Alternate Day Dosing

SUMMARY:
Iron is very important for our body and performs vital tasks. Iron deficiency is a worldwide health problem. The prevalence of anemia in women of reproductive age in Southeast Asia is estimated to be 46.6% in 2019, with iron deficiency being one of the main reasons for anemia. There are different approaches to treat iron deficiency. One of them is the use of iron supplements. Recommended iron supplement treatments today often differ in dose, regimen and length. Experts recommend a dose of 80-200 mg of iron taken either daily or on several days per week, depending on the severity of the iron deficiency (with or without anemia). From certain guidelines lower amounts of iron are also recommended, as this could lead to fewer side effects.Previous studies have shown that both daily and multiple days per week administration can be effective in treating iron deficiency. Recently, several successive iron supplementation studies in Zurich showed that 24 h after ingestion of an oral dose of >60mg iron, the absorption of iron in the body is impaired. In addition it was measured that iron supplements taken only every other day instead of every day are absorbed about 30-50% better and have fewer side effects. Little is known about the long-term effect of this alternating regimen on iron status and side effects.With this 6-months study in the Philippines, the investigators want to compare two different supplementation regimens with oral iron to see if there is any difference in the iron status, intestinal inflammation levels, and side effects, and therefore if it would be better to take the iron supplements every 2 days instead of daily.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 45 years old,
* SF levels <25 µg/L,
* Hb levels 11-15.5 g/dL
* Normal Body Mass Index (18.5-25 kg/m2),
* In possession of a mobile phone on which the study app can be loaded
* Signed informed consent

Exclusion Criteria:

* Elevated CRP > 5 mg/L
* Any metabolic, gastrointestinal, kidney or chronic disease such as diabetes, renal failure, hepatic dysfunction, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement) affecting iron metabolism,
* Use of medication which may interfere with iron absorption, gut physiology and iron metabolism
* Consumption of iron supplements within 2 weeks prior to study start and of additional iron supplements during the study period
* Difficulties with blood sampling,
* Known hypersensitivity or allergy to iron or placebo capsules in the given amount (ferrous sulfate, mannitol, silica)
* Pregnancy, breastfeeding
* Known or suspected non-compliance, drug or alcohol abuse
* Cigarette smokers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Woman
Enrollment: 22 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2022-11-19 (Actual)

PRIMARY OUTCOMES:
Serum Ferritin (SF) | Day 93
  in consecutive day group
Serum Ferritin (SF) | Day 186
  in alternate day group
Event rate of GI side effects | Day 90
  in consecutive day group
Event rate of GI side effects | Day 183
  in alternate day group

SECONDARY OUTCOMES:
Hemoglobin (Hb) | Day 0
Hemoglobin (Hb) | Day 46
Hemoglobin (Hb) | Day 93
Hemoglobin (Hb) | Day 139
Hemoglobin (Hb) | Day 183
Serum Ferritin (SF) | Day 0
Serum Ferritin (SF) | Day 46
Serum Ferritin (SF) | Day 93
Serum Ferritin (SF) | Day 139
Serum Ferritin (SF) | Day 186
Serum Transferrin Receptor (sTfR) | Day 0
Serum Transferrin Receptor (sTfR) | Day 46
Serum Transferrin Receptor (sTfR) | Day 93
Serum Transferrin Receptor (sTfR) | Day 139
Serum Transferrin Receptor (sTfR) | Day 186
Total iron binding capacity (TIBC) | Day 0
Total iron binding capacity (TIBC) | Day 93
Total iron binding capacity (TIBC) | Day 186
Serum Iron (SFe) | Day 0
Serum Iron (SFe) | Day 93
Serum Iron (SFe) | Day 186
C-Reactive Protein (CRP) | Day 0
C-Reactive Protein (CRP) | Day 46
C-Reactive Protein (CRP) | Day 93
C-Reactive Protein (CRP) | Day 139
C-Reactive Protein (CRP) | Day 186
Alpha-1-acid Glycoprotein (AGP) | Day 0
Alpha-1-acid Glycoprotein (AGP) | Day 46
Alpha-1-acid Glycoprotein (AGP) | Day 93
Alpha-1-acid Glycoprotein (AGP) | Day 139
Alpha-1-acid Glycoprotein (AGP) | Day 186
Intestinal Fatty Acid-binding Protein (I-FABP) | Day 0
Intestinal Fatty Acid-binding Protein (I-FABP) | Day 90
Intestinal Fatty Acid-binding Protein (I-FABP) | Day 183
Calprotectin | Day 0
Calprotectin | Day 90
Calprotectin | Day 183
Hepcidin | Day 0
Hepcidin | Day 46
Hepcidin | Day 90
Hepcidin | Day 139
Hepcidin | Day 183
Event rate of GI side effects | Day 90
Event rate of GI side effects | Day 183
Incidence of GI side effects | Day 90
Incidence of GI side effects | Day 183
Event proportion of GI side effects | Day 90
Event proportion of GI side effects | Day 183
Severity of GI side effects | Day 90
  5 different side effects (nausea, stomach pain, constipation, diarrhea, bloating) are reported if they occur in a study app and rated "mild" or "severe", according to their judgement.
Severity of GI side effects | Day 183
  5 different side effects (nausea, stomach pain, constipation, diarrhea, bloating) are reported if they occur in a study app and rated "mild" or "severe", according to their judgement.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Santo Tomas Hospital, Manila, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: No